CLINICAL TRIAL: NCT06151054
Title: Relationship Between Aortic Parietal Inflammation on 18F-FDG PET Scan and Arterial Stiffness as a Function of Age
Acronym: RAIPAo
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pierre Yves MARIE, professor, Central Hospital, Nancy, France
Other Study IDs: 2022PI141
Record Dates: First submitted 2022-09-08; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Arterial Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measure of aortic inflammation — Standard Uptake Value (SUV) measures of aortic wall

SUMMARY:
Show that there is a relationship between arterial stiffness and aortic parietal inflammation and that this relationship is different in the three age groups with aortic parietal inflammation occurring earlier than arterial stiffness.

DETAILED DESCRIPTION:
In the literature, a relationship has been demonstrated between local inflammation in the aortic wall and increased arterial stiffness. Arterial stiffness is commonly represented by pulse wave velocity (PWV) measured using an applanation tonometer. It would seem that this parietal inflammation precedes arterial stiffness and consequently, arterial hypertension . Arterial stiffness is an important factor of cardiovascular morbidity and mortality and therefore represents a major public health interest in prevention in the face of the continuous aging of our population . This study will consist in studying on a population divided into three age groups, less than 40 years old, 40 to 60 years old and more than 60 years old, the relationship between thoracic aortic parietal inflammation evaluated using the Standard Uptake Value parameters (SUV) and Hounsfield units (HU) measured on 18F-FDG PET/CT scans performed between 09/04/2018 and 11/06/2020 and arterial stiffness parameters. We will seek to show that there is a relationship between arterial stiffness and aortic parietal inflammation and that this relationship is different in the three age groups with aortic parietal inflammation occurring earlier than arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent whole-body 18F-FDG PET/CT included in the PACTEP study
* Patient with an assessment of arterial stiffness by applanation tonometer

Exclusion Criteria:

* patients without an assessment of arterial stiffness by applanation tonometer

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent whole-body 18F-FDG PET/CT included in the PACTEP study and in this context, who had an assessment of arterial stiffness by applanation tonometer
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
to etablish a relationship inflammation of aortic wall and arterial stiffness | 1 day
  Standard Uptake Value

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie HUE, MSc, Study Director — CHRU Nancy
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France